CLINICAL TRIAL: NCT03502291
Title: The Effect of Live Attenuated Inactivated Influenza Vaccine on Experimental Human Pneumococcal Carriage Study
Acronym: LAIV/EHPC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: Sponsor GmbH (Other); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 4896
Record Dates: First submitted 2016-10-18; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2016-05

CONDITIONS: Pneumonia; Influenza, Human
Keywords: Human challenge models; Immunity; Streptococcus pneumoniae; Live Attenuated Influenza Vaccine
MeSH Terms: conditions — Pneumonia; Influenza, Human | interventions — Vaccination; FluMist

STUDY DESIGN:
Intervention Model Description: DBRCT performed as two studies over two flu seasons. 2 arms to each study.
Who Masked: Participant, Investigator
Masking Description: Physical blind folds worn by participant. Unblinded research nurses to deliver the vaccines
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Study One: LAIV + Inoculation (Active Comparator): LAIV Nasal Spray: Inoculation (FLUMIST or FLUENZ) plus intramuscular placebo then inoculation with pneumococci bacteria
  Interventions: Biological: Study one: LAIV + Inoculation
- Study One: Placebo + inoculation (Placebo Comparator): Quadrivalent Inactivated Influenza Vaccine Intramuscular (Fluarix Tetra) plus nasal placebo then inoculation with pneumococci bacterial
  Interventions: Biological: Study one: Placebo + Inoculation
- Study Two: Inoculation + LAIV (Active Comparator): Inoculation with pneumococci bacteria then Live attenuated Influenza Vaccine Nasal Spray (FLUMIST or FLUENZ) plus intramuscular placebo
  Interventions: Biological: Study two: Inoculation + LAIV
- Study Two: Inoculation + placebo (Placebo Comparator): Inoculation with pneumococci bacteria then Quadrivalent Inactivated Influenza Vaccine Intramuscular (Fluarix Tetra) plus nasal placebo
  Interventions: Biological: Study two: Inoculation + placebo

INTERVENTIONS:
Biological: Study one: LAIV + Inoculation — Pneumococci bacteria nasal inoculation following vaccination with LAIV and intramuscular placebo
  Other Names: FLUMIST or FLUENZ AstraZeneca
  Arms: Study One: LAIV + Inoculation
Biological: Study one: Placebo + Inoculation — Pneumococci bacteria nasal inoculation following vaccination QIV with nasal placebo spray
  Other Names: Fluarix Tetra GlaxoSmithKline
  Arms: Study One: Placebo + inoculation
Biological: Study two: Inoculation + LAIV — Pneumococci bacteria nasal inoculation prior to vaccination with LAIV and intramuscular placebo
  Other Names: FLUMIST or FLUENZ AstraZeneca
  Arms: Study Two: Inoculation + LAIV
Biological: Study two: Inoculation + placebo — Pneumococci bacteria nasal inoculation prior to vaccination QIV with nasal placebo
  Other Names: Fluarix Tetra GlaxoSmithKline
  Arms: Study Two: Inoculation + placebo

SUMMARY:
The investigators are interested in examining the effect of the Live Attenuated Influenza (flu) Vaccine (LAIV) upon nasal carriage of bacteria called Streptococcus pneumoniae (also known as pneumococcus). The nasal spray is a live attenuated vaccine which means that it has weakened virus that does not cause disease. This vaccine is licenced in the United Kingdom for children and adolescents from 2 to 18 years of age.

Pneumococcus can commonly be found harmlessly inhabiting the nose where it does not cause any problem (pneumococcal colonisation). About 10% of adults carry pneumococcus at any one time, and almost all adults experience an episode of carriage at least once per year. Carriage acts as a natural vaccine, boosting immunity against pneumococcal infection in adults and children.

During influenza there is an increase in the burden of pneumococcal pneumonia. We have studied the effects of pneumococcus for many years and have developed a programme in which we can nasally inoculate healthy participants with a dose of pneumococcus and achieve a reproducible carriage rate. The investigators would now like to use this model to investigate the effects of the nasal influenza vaccine upon pneumococcal carriage and to better understand how influenza infections lead to increased susceptibility to pneumonia.

Pneumococcal disease in young adults is rare - less than 10 cases per 100,000 people per year. When pneumococcus does cause problems, usually in young children or elderly people, it can be very serious as it is responsible for diseases such as pneumonia, sepsis and meningitis, which kill millions of children around the world each year.

DETAILED DESCRIPTION:
Secondary bacterial infections such as pneumococcal pneumonia are a leading cause of death during influenza endemics. Individuals recently infected with influenza become more susceptible to pneumonia, an effect associated with increased density of pneumococcal carriage in the nose and uncontrolled inflammatory immunological responses. The interaction of influenza virus and pneumococcus has been known and well documented. Recent works have shown that the Live Attenuated Influenza Vaccine (LAIV) enhances pneumococcal carriage in murine models. These results highlighted the potential effect of mass immunization of children with LAIV on pneumococcal carriage. Increased carriage could lead to increased pneumococcal disease in LAIV-vaccinated individuals as well as increased bacterial transmission within the population. LAIV has been licensed for use in children since 2011 in Europe, and has been increasingly administered in children and adults in the USA. There is an urgent need for a clinical trial that will determine the effect of LAIV on pneumococcal carriage dynamics.

The investigators have developed a safe and reproducible experimental human pneumococcal carriage (EHPC) model. The investigators will use EHPC to define the effect of antecedent and concurrent LAIV on pneumococcal carriage acquisition, density and duration. The investigators will perform two double - blinded Randomised Controlled Trials (RCT) to compare LAIV with Quadrivalent Inactivated Influenza Vaccine (QIV). The investigators will compare clinical symptoms, pneumococcal carriage density and duration associated with both vaccines administered antecedent to or concurrently with EHPC inoculation. Changes in the nasopharyngeal microbiome, inflammatory responses in the nasal mucosal and lung cellular immunity associated with influenza virus and pneumococcus interaction will be investigated. This project may provide some reassurance regarding the impact of mass immunization with LAIV on carriage or, if carriage is increased, will provide knowledge of how a natural carriage episode might develop into pneumonia in susceptible subjects during pandemic influenza.

ELIGIBILITY:
Inclusion Criteria:

* have capacity to give informed consent
* aged 18-50 yrs - ages chosen to minimise the risk of pneumococcal infection
* speak fluent English- to ensure a comprehensive understanding of the research project and their proposed involvement, in order to minimise any communication issues to maximise participant safety.

Exclusion Criteria:

* currently involved in another study unless observational or in follow-up phase (non-interventional)
* received any influenza vaccine in the last 2 years

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 324 (Actual)
Dates: Start 2015-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Detection of pneumococcal bacteria in the nasal wash sample | within 6 weeks of inoculation per patient
  Primary outcome: detection of pneumococcal bacteria in the nasal wash sample at any time point after inoculation by classical microbiology. 130 participants will complete the study (65 in each arm) to achieve 80% power to detect 50% increase in colonisation rates induced by antecedent LAIV compared to control

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Rylance, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Royal Liverpool Hospital, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitsi E, Reine J, Urban BC, Solorzano C, Nikolaou E, Hyder-Wright AD, Pojar S, Howard A, Hitchins L, Glynn S, Farrar MC, Liatsikos K, Collins AM, Walker NF, Hill HC, German EL, Cheliotis KS, Byrne RL, Williams CT, Cubas-Atienzar AI, Fletcher TE, Adams ER, Draper SJ, Pulido D, Beavon R, Theilacker C, Begier E, Jodar L, Gessner BD, Ferreira DM. Streptococcus pneumoniae colonization associates with impaired adaptive immune responses against SARS-CoV-2. J Clin Invest. 2022 Apr 1;132(7):e157124. doi: 10.1172/JCI157124. PMID 35139037